CLINICAL TRIAL: NCT04572828
Title: Effectiveness of Paracervical Block in Endometrial Sampling Procedures for Pain Control: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Paracervical Block in Endometrial Sampling Procedures for Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-6.1T/67
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Office-based Endometrial Sampling Procedures
MeSH Terms: interventions — Anesthesia, Obstetrical; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Waiting 1 Minute After Paracervical Block (Active Comparator)
  Interventions: Procedure: Paracervical Block
- Group 2: Waiting 3 Minute After Paracervical Block (Active Comparator)
  Interventions: Procedure: Paracervical Block
- Group 3: Control Group (Placebo Comparator)
  Interventions: Procedure: The capped needle
- Group 4: Waiting 60 Minute After Taking Oral NSAIDs (Active Comparator)
  Interventions: Drug: 550 mg Naproxen Sodium 60 minutes before the procedure

INTERVENTIONS:
Procedure: Paracervical Block — Two-point (at 4 and 8 o'clock only) technique will be used for paracervical block for Group 1: Waiting 1 Minute After Paracervical Block and Group 2: Waiting 3 Minute After Paracervical Block. For these groups 10 ml 2% Prilocaine (VEM İlac, Tekirdag, Turkey) will be injected for each side approximately 10 mm into the cervical stroma at the cervico-vaginal junction with a 22- gauge hypodermic needle.
  Other Names: 550 mg Naproxen Sodium 60 minutes before the procedure.
  Arms: Group 1: Waiting 1 Minute After Paracervical Block; Group 2: Waiting 3 Minute After Paracervical Block
Drug: 550 mg Naproxen Sodium 60 minutes before the procedure — 550 mg Naproxen Sodium (Abdi Ibrahim, Turkey) will be given to participants in the Group 4, 60 minutes before the procedure.
  Arms: Group 4: Waiting 60 Minute After Taking Oral NSAIDs
Procedure: The capped needle — The capped needle model will be employed for Group 3: Control Group. After cervical and vaginal preparation with povidone iodine a capped needle will be touched the cervico-vaginal junction at 4 and 8 o'clock.
  Arms: Group 3: Control Group

SUMMARY:
Office-based endometrial procedures are preferred over diagnostic dilation and curettage, nowadays. Paracervical block is single-shot nerve block that involve a one-time injection of local anesthetic adjacent to the utero-vaginal nerve plexus. Block provides analgesia during cervical pass of sampling device or manipulation of cervix. The paracervical block seems to work within few minutes after injection, but the optimal waiting time between injection and procedure is not known. In this randomized controlled study, it was aimed to determine the effect of waiting time of 1 minute and 3 minutes after paracervical block in endometrial sampling procedures using Pipelle cannula in terms of pain during and after the endometrial sampling and to compare with NSAIDs taken before the procedure.

DETAILED DESCRIPTION:
120 participants who will undergo endometrial biopsy due to abnormal uterine bleeding will be enrolled in the study. The research will be conducted in 4 branches. These branches are Group 1: Waiting 1 Minute After Paracervical Block, Group 2: Waiting 3 Minute After Paracervical Block, Group 3: Control Group and Group 4: Waiting 60 Minute After Taking Oral NSAIDs. Thirty patients will be included in each group using power analysis of clinical studies in which endometrial biopsy techniques and pain comparisons were performed before [Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018;132(3):575-582.].

Pregnancy, pelvic infections, heavy bleeding disorders and NSAID allergy are the exclusion criteria.

In the study, the success of analgesic methods to be used for endometrial biopsy during and 30 minutes after the procedure will be compared. These methods include waiting 1 minute after the paracervical block is performed, waiting 3 minutes after the paracervical block is performed, and taking oral NSAIDs one hour before the procedure. All arms will be included 30 participants and control group with 30 participants is formed. The Numeric Pain Rating Scale (NPRS) system will be used for each case for pain during the procedure and 30 minutes after the procedure. According to this system, the fact that the participant have no pain will be evaluated as "0" point and having the most severe pain she can experience is "10" points.

Before procedure the cervix and vaginal vault will be prepared with povidone iodine. A vaginal speculum will be used for optimal exposure and manipulation of cervix. All procedures will be performed without grasping the cervix with a tenaculum. Two-point (at 4 and 8 o'clock only) technique will be used for paracervical block for Group 1: Waiting 1 Minute After Paracervical Block and Group 2: Waiting 3 Minute After Paracervical Block. For these groups 10 ml 2% Prilocaine (VEM İlac, Tekirdag, Turkey) will be injected for each side approximately 10 mm into the cervical stroma at the cervico-vaginal junction with a 22- gauge hypodermic needle. The capped needle model will be employed for Group 3: Control Group. After cervical and vaginal preparation with povidone iodine a capped needle will be touched the cervico-vaginal junction at 4 and 8 o'clock. 550 mg Naproxen Sodium (Abdi Ibrahim, Turkey) will be given to participants in the Group 4, 60 minutes before the procedure.

For all procedures, low pressure sampling device (Pipelle Cannula, Medbar Medical Equipment Inc.)will be inserted to the cavity and endometrial samples will be obtained using a corkscrew rotation combined with a repeating cephalic-caudal motion. The procedure will be repeated twice in each case to ensure standardization. All endometrial biopsies will be performed by the same operator.

NPRS system will be explained to all groups after the procedure and the pain during the procedure will be requested to be graded. Thirty minutes after the procedure, the participants will be asked to rate current pain according to the NPRS system.

The study was approved by institutional ethics committee. Written informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding

Exclusion Criteria:

* Pregnancy
* Pelvic infections
* Heavy bleeding disorders
* NSAID allergy

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale 0 | Baseline (0 minute)
  The Numeric Pain Rating Scale (NPRS) system will be used for each case for pain during the procedure. According to this system, the fact that the participant has no pain is evaluated as "0" point and having the most severe pain she could experience is "10" points.
The Numeric Pain Rating Scale 30 | 30 minutes
  The Numeric Pain Rating Scale (NPRS) system will be used for each case for pain 30 minutes after procedure. According to this system, the fact that the participant has no pain is evaluated as "0" point and having the most severe pain she could experience is "10" points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol